CLINICAL TRIAL: NCT02969291
Title: A Home-Based Study to Enhance Activity in Breast Cancer Survivors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Baystate Medical Center (Other)
Collaborators: University of Massachusetts, Amherst (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 776553-5
Record Dates: First submitted 2016-11-02; First posted 2016-11-21 (Estimated); Last update posted 2019-07-17 (Actual); Status verified 2019-07

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Reduced Sedentary Time Intervention (Other): Reduced Sedentary Time Intervention (RSTI)
  Interventions: Behavioral: Reduced Sedentary Time Intervention (RSTI)

INTERVENTIONS:
Behavioral: Reduced Sedentary Time Intervention (RSTI) — Following 7 days of baseline activity monitoring a study investigator will download the information from the monitor, evaluate the periods of sedentary behavior and create a tailored RSTI for each participant. For example, the investigator may notice a long stretch of sitting in the evening following a meal and identify several exercises that can be done indoors during that time, or if the participant is amiable to walking breaks and a period after work is identified the investigator might suggest the appropriate walking activity at that time. This program has been successful in sedentary overweight office workers and investigators will use similar techniques.

SUMMARY:
There is a well-documented association between physical activity & risk for breast cancer development and recurrence. It is known that exercise interventions have been effective at increasing physical activity levels in breast cancer survivors. Knowing that breast cancer survivors are less active than non-cancer patients, a less active lifestyle places them at risk of obesity and poor overall health, which in turn also increases risk of cancer and cancer recurrence. Not all the reasons for the risk reduction are clear, however it is known that hormones and other inflammatory markers play a role.

This study has three goals:

1. To investigate the feasibility of a home intervention designed to reduce sedentary behavior.
2. Describe the effects of the intervention on levels of sedentary behavior, physical activity, and symptoms.
3. Assess cost of the intervention.

DETAILED DESCRIPTION:
There is a well-documented association between physical activity and risk for breast cancer development and recurrence. Exercise training interventions have been effective at increasing physical activity levels in breast cancer survivors, however they require 1) a large degree of patient initiative to achieve positive health outcomes associated with sustained behavioral change and 2) facilities and oversight that may be prohibitive in a clinical setting. Although most activity-based research to date has focused on increasing levels of moderate to vigorous physical activity (MVPA) for breast cancer survivors, large epidemiological studies suggest that breast cancer survivors are also more sedentary when compared to non-cancer controls. A recent meta-analysis of controlled intervention trials designed to promote physical activity among sedentary cancer survivors found that none of the trials within the scope of the review succeeded in achieving 75% or better adherence to prescribed exercise guidelines, leading the authors to question whether shifting the target of intervention from MVPA to reductions in sedentary time might be a more realistic goal. Recent research suggests that interventions designed to reduce sedentary time in breast cancer survivors have the potential to yield clinically meaningful health benefits, especially for individuals at higher risk for sedentary behaviors, however the optimal method of intervention is not clear.

Aim 1: Feasibility of the intervention Assess the feasibility of an intervention designed to reduce sedentary behavior in breast cancer survivors. The behavioral intervention will involve the review of a 7-day baseline snapshot of sedentary behavior and physical activity patterns, combined with tailored activity prompts described over the following 6 weeks.

Aim 2: Effects of the intervention Aim 2a: Describe a preliminary range of effect sizes of the intervention on levels of sedentary behavior, physical activity and symptoms of cancer survivorship (e.g. cancer related fatigue).

Aim 2b: Evaluate the relationship between change in sedentary behavior and change in cancer-relevant outcomes, such as fatigue and biomarkers of cancer recurrence (e.g. IGF-1, Leptin), following the reduced sedentary time intervention.

Aim 3: Assessment of intervention components Aim 3a: Quantitatively assess overall cost of the intervention and its individual components, dose delivered and dose received by intervention participants Aim 3b: Quantitatively describe intervention participants' perspectives on the impact of the individual intervention components, including which components appeared most useful for reducing sedentary time.

ELIGIBILITY:
Inclusion Criteria:

* Stage I-III breast cancer survivors 20-80 who have completed primary treatment (surgery, radiation and/or chemotherapy) greater than 6 months but less than 5 years ago. Patients may be on adjuvant hormonal therapy
* BMI > 25 (overweight or class I/II obese)
* Not meeting current guidelines for regular exercise as defined by less than 150 minutes a week of moderate to vigorous physical activity
* No gain or loss of >10% body weight over the prior 6 months.

Exclusion Criteria:

* Known diabetes
* Known coronary artery disease
* Pregnancy
* Any injury that would limit mobility or require use of assisted mobility devices
* Weight gain or loss of >10% body weight over the prior 6 months
* Greater than 150 minutes a week of moderate to vigorous physical activity
* Inability to provide informed consent
* Non-english speaking

Ages: 20 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2016-10; Primary Completion 2018-10 (Actual); Study Completion 2018-10 (Actual)

PRIMARY OUTCOMES:
Sedentary Time | 8 weeks
  Change in minutes/day of sedentary time as recorded by ActivPal in all 25 participants pre and post intervention.

SECONDARY OUTCOMES:
Activity Level | 8 weeks
  Change in Activity level as recorded by Actigraph monitor in all 25 participants
Glucose | 8 weeks
  Change in fasting glucose ( mmol/L)in all 25 participants
Insulin | 8 weeks
  Change in insulin (pmol/L) in all 25 participants
Total cholesterol | 8 weeks
  Change in total cholesterol (mmol) in all 25 participants
High density lipoprotien cholesterol | 8 weeks
  Change in high density lipoprotein cholesterol (mmol) in all 25 participants
Triglyceride | 8 weeks
  Change in triglycerides (mmol) in all 25 participants
Body Mass Index | 8 weeks
  Change in Body Mass Index (kg/m2) in all 25 participants
Waist Circumference | 8 weeks
  Change in waist circumference in cm in all 25 participants
Systolic Blood pressure | 8 weeks
  Change in systolic blood pressure measured in mmHg in all 25 participants
Diastolic Blood pressure | 8 weeks
  Change in diastolic blood pressure measured in mmHg in all 25 participants
Cancer-related fatigue measured by change in PROMIS short form 8a in all 25 participants | 8 weeks
Cancer-related fatigue as measured by change in Visual Analog scale in all 25 participants | 8 weeks
Sedentary behavior self -efficacy | 8 weeks
  Change in Sedentary Behavior Self-Efficacy Scale (modified from BARSE) in all 25 participants
Change in EORTC-QLQ-C30 scores in all 25 participants | 8 weeks
Assessment of Intervention | 8 weeks
  Change in Assessment of Intervention questions on a scale of 1-5 in all 25 participants

CONTACTS AND LOCATIONS:
Overall Officials: Grace Makari-Judson, MD, Principal Investigator — Baystate Medical Center
Locations (1):
- Baystate Medical Center, Springfield, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Undecided